CLINICAL TRIAL: NCT04690946
Title: Randomized Controlled Study Comparing the Therapeutic Effect and Change Processes in Cognitive Behavioral Therapy and Emotion-Focused Therapy for Depression
Brief Title: Comparing Effect and Change Processes in Cognitive Behavioral Therapy and Emotion-Focused Therapy for Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institutt for Psykologisk Radgivning (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPR
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Emotion-Focused Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): 14-18 sessions of psychotherapy according to principles of Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Emotion-Focused Therapy (Active Comparator): 14-18 sessions of psychotherapy according to principles of Emotion Focused Therapy
  Interventions: Behavioral: Emotion-Focused Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 14-18 sessions of CBT
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Emotion-Focused Therapy — 14-18 sessions of EFT
  Other Names: EFT
  Arms: Emotion-Focused Therapy

SUMMARY:
Depression is a common mental illness which is costly for both society and for those affected. There is a need for effective treatments of depression and there is a need to make sure that the treatments that are given are based on scientific findings. In this study the investigators want to examine and compare two common treatment models for depression - Cognitive Behavioral Therapy and Emotion-Focused Therapy. The investigators want to investigate what characterizes these treatments when they are successful, and seek to better understand what it is like for patients to receive these treatments. Also, the investigators will investigate the experience of patients who abruptly discontinue treatment. To investigate these questions, self-report measures, interviews and analysis of session recordings will be used.

DETAILED DESCRIPTION:
Depression is a widespread mental disorder which can result in severe impairment and reduced quality of life for those affected. Cognitive behavioral therapy (CBT) is the approach with strongest empirical support, and is often recommended as treatment for depression, as in the NICE Guidelines for Depression from 2009. However, research indicates that not all patients respond to CBT, indicating a need to expand the range of available evidence-based psychotherapies, and mapping the mechanisms of change in existing treatments.

Emotion focused therapy (EFT) is one promising treatment for depression with empirical support for its efficacy. A previous study found equal outcome in CBT and Process-Experiential treatment/EFT for depression, but more studies are needed to replicate these findings across cultural contexts. The main aim of this study is to investigate whether there are significant differences in the therapeutic effect of EFT compared to that of CBT for patients with moderate and major depressive disorder in a Norwegian outpatient setting.

Although several psychotherapeutic approaches have shown efficacy in the treatment of depression, no psychotherapeutic interventions is beneficial for all patients. There is a need for research that investigates what treatments works for whom, based on patient characteristics and preferences. The present study will investigate whether patient characteristics moderate treatment outcome, both within and between treatment conditions. In addition, qualitative interviews will be conducted to get a deeper understanding of what clients find helpful and challenging within the CBT and EFT condition, and to explore the experience of patients who drop-out of the treatment process.

In order to further develop psychotherapeutic treatments and increase their effectiveness, there is a need to identify processes that are related to good and poor outcome. Process-outcome studies are commonly used for this purpose. The present study will investigate and compare characteristics of psychotherapy processes in both the CBT and EFT conditions and how these are related to outcome.

Study design and Method

The study will be conducted as a randomized controlled trial (RCT) in order to compare the efficacy of EFT to CBT. RCT's are considered the gold standard for efficacy studies. Participants will be recruited from the Norwegian mental health program "Return to work", a publicly funded treatment program where patients with common mental health issues receives outpatient psychotherapeutic treatment to reduce and prevent sick leave.

The present study will address the following research hypothesis and questions:

1. EFT and CBT will not result in significantly different outcome in the treatment of patients with moderate and major depressive disorder.
2. Patient characteristics (severity of depression, adverse childhood experiences and clients' initial ability to make sense of their experience) will moderate treatment outcome for both conditions.
3. Will therapeutic processes (therapeutic alliance, therapist empathy, clients' ability to make sense of their experience and emotional processing) mediate treatment outcome equally for both conditions?
4. What do patients in both conditions describe as helpful and unhelpful aspects of treatment?
5. How do patients in both conditions describe their own change or lack or change after treatment?
6. How do patients that choose to drop out of treatment describe the processes leading to that decision?

ELIGIBILITY:
Inclusion Criteria:

- Moderate or major depressive episode as primary diagnosis

Exclusion Criteria:

* Serious mental illness (schizophrenia, severe bipolar disorder, recent or current psychotic episode) or intellectual disability.
* Severe alcohol or drug abuse, last 12 months.
* Suicidality last 6 months
* Severe medical issues
* If the participant is on antidepressive medication, the dosage must have been stable for more than 4 weeks, and the participant must consent to staying on the same dosage for the duration of the treatment.
* The participant is currently in another treatment for depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory from session to session | 1 week before treatment startup, 1 day after each therapy session, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of depressive symptoms, ranging from minimum 0 and maximum 63. Higher scores suggests worse outcome.

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of anxiety symptoms, ranging from minimum 0 and maximum 63. Higher scores suggests worse outcome.
Change in Repetitive Eating Questionnaire | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of symptoms related to eating disorders, average scores, minimum 0, maximum 6, higher score indicates worse outcome.
Change in Inventory of Interpersonal problems | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of interpersonal difficulties, average scores minimum 0, maximum 4. Higher score suggests worse outcome.
Change in The Acceptance and Action Questionnaire from session to session | 1 week before treatment startup, 1 day after each therapy session, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of psychological flexibility, average scores minimum 1, maximum 7. Higher score suggests worse outcome.
Change in Emotion Approach Coping Scale | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of emotional processing ability, average scores minimum 1, maximum 4. Higher score suggests better outcome.
Change in Penn State Worry Questionaire | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of rumination and cognitive processing, total scores minimum 16, maximum 80. Higher score suggests worse outcome.
Change in Self-Compassion Scale | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of self-relating, average scores, minimum 1, maximum 5, higher scores suggests better outcome.
Change in Quality of life questionnaire | 1 week before treatment startup, within 1 week after treatment, 3 month follow up, 6 month follow up, 12 months follow up
  Self-report measure of quality of life, average scores, minimum 1, maximum 5, higher scores indicate better outcome.
Change in Working Alliance Inventory - short version | 1 day after 1st through 14th therapy session.
  Self report measure on experience of therapeutic alliance, average scores, minimum 1, maximum 7, higher scores suggests better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Reidar Stiegler, PhD, Principal Investigator — Institute for Psychological Counselling
Locations (1):
- Institutt for Psykologisk rådgivning, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimidjian S, Hollon SD. How would we know if psychotherapy were harmful? Am Psychol. 2010 Jan;65(1):21-33. doi: 10.1037/a0017299. PMID 20063907
- [Background] Blatt SJ, Luyten P. A structural-developmental psychodynamic approach to psychopathology: two polarities of experience across the life span. Dev Psychopathol. 2009 Summer;21(3):793-814. doi: 10.1017/S0954579409000431. PMID 19583884
- [Background] Elliott R. Psychotherapy change process research: realizing the promise. Psychother Res. 2010 Mar;20(2):123-35. doi: 10.1080/10503300903470743. PMID 20099202
- [Background] Goldman, R. N., Greenberg, L. S., & Angus, L. (2006). The effects of adding emotion-focused interventions to the client-centered relationship conditions in the treatment of depression. Psychotherapy Research, 16(5), 537-549.
- [Background] Watson JC, Gordon LB, Stermac L, Kalogerakos F, Steckley P. Comparing the effectiveness of process-experiential with cognitive-behavioral psychotherapy in the treatment of depression. J Consult Clin Psychol. 2003 Aug;71(4):773-81. doi: 10.1037/0022-006x.71.4.773. PMID 12924682
- [Background] Greenberg, L & Watson, J. (1998). Experiential Therapy of Depression: Differential Effects of ClientCentered Relationship Conditions and Process Experiential Interventions, Psychotherapy Research, 8:2, 210-224.
- [Background] Kazdin AE. Understanding how and why psychotherapy leads to change. Psychother Res. 2009 Jul;19(4-5):418-28. doi: 10.1080/10503300802448899. PMID 19034715
- [Background] Kazdin AE. Evidence-based treatment research: Advances, limitations, and next steps. Am Psychol. 2011 Nov;66(8):685-698. doi: 10.1037/a0024975. PMID 22082384
- [Background] Kendall JM. Designing a research project: randomised controlled trials and their principles. Emerg Med J. 2003 Mar;20(2):164-8. doi: 10.1136/emj.20.2.164. No abstract available. PMID 12642531
- [Background] Lambert, M. J. (2011). What have we learned about treatment failure in empirically supported treatments? Some suggestions for practice. Cognitive and Behavioral Practice, 18(3), 413-420.
- [Background] What have we learned about treatment failure in empirically supported treatments
- [Background] NICE (2009a). Depression: Treatment and Management of Depression in Adults. Clinical Guideline 90. London: National Institute for Health and Clinical Excellence. Available at www.nice.org.uk
- [Background] Nilsson, T., Svensson, M., Sandell, R. & Clinton, D. (2007). Patients' experiences of change in cognitive-behavioral therapy and psychodynamic therapy: a qualitative comparative study. Psychotherapy Research, 17:5, 553-566.
- [Background] Rice, L. N., & Greenberg, L. S. (Eds.). (1984). Patterns of change: Intensive analysis of psychotherapy process. Guilford Press.
- [Background] Roth, A & Fonagy, P (1996) What works for whom? New York: Guilford Press
- [Background] Watson JC. Mapping patterns of change in emotion-focused psychotherapy: Implications for theory, research, practice, and training. Psychother Res. 2018 May;28(3):389-405. doi: 10.1080/10503307.2018.1435920. Epub 2018 Feb 21. PMID 29466928
- [Derived] Aardal H, Schanche E, Hjeltnes A, Danielsen YS. Cognitive behavioral therapy and emotion-focused therapy for depression in a routine care setting: A randomized controlled pilot trial. Psychother Res. 2025 Oct 1:1-15. doi: 10.1080/10503307.2025.2560935. Online ahead of print. PMID 41031587

DOCUMENTS (1):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04690946/Prot_001.pdf